CLINICAL TRIAL: NCT02053051
Title: Clinical Assessment of an Advanced Bolus Calculator for Type 1 Diabetes (ABC4D)
Brief Title: Advanced Bolus Calculator for Type 1 Diabetes (ABC4D)
Acronym: ABC4D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13SM0091
Record Dates: First submitted 2014-01-22; First posted 2014-02-03 (Estimated); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Advanced Bolus Calculator
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 4: Intervention (ABC4D) (Experimental): Advanced Bolus Calculator for Type Diabetes (ABC4D)
  Interventions: Device: ABC4D
- Phase 4 Control: Standard bolus calculator (Active Comparator): Standard bolus calculator
  Interventions: Device: Standard bolus calculator

INTERVENTIONS:
Device: ABC4D — Advanced Bolus Calculator for Type 1 Diabetes (ABC4D) to calculate pre-meal insulin boluses
  Arms: Phase 4: Intervention (ABC4D)
Device: Standard bolus calculator
  Arms: Phase 4 Control: Standard bolus calculator

SUMMARY:
This study aims to assess the safety and efficacy of a novel advanced bolus calculator in subjects with Type 1 diabetes. Insulin bolus calculators have been developed to aid insulin dose adjustment and existing standard insulin bolus calculator consist of a simple algorithm that requires five subject-specific parameters as input to generate a recommended bolus insulin dose:

* current blood glucose (mmol/L)
* target blood glucose (mmol/L)
* insulin-to-carbohydrate ratio (grams of carbohydrate per 1 unit of insulin)
* total grams of carbohydrate in meals
* insulin sensitivity factor (reduction in glucose per 1 unit of insulin)

DETAILED DESCRIPTION:
The Diabetes Technology team at Imperial College have developed a novel advanced bolus calculator. The complete integrated system consists of a commercially available smartphone that holds the novel advanced algorithm. The system requires regular updates of cases derived from retrospective blinded continuous glucose monitoring data and for this a commercially available glucose sensor will be used. Each new case includes information about the problem (e.g. capillary blood glucose, meal information and physical exercise), solution (recommended insulin dose) and outcome (blood glucose following a meal). The novel decision support algorithm is based on case-based reasoning (CBR). CBR is an artificial intelligence technique that tries to solve newly encountered problems by applying the solutions learned from solved problems encountered in the past.

The end-product is therefore a subject specific insulin bolus calculator that continues to improve with time. The project utilises commercially available glucose sensors and smartphones (iPhone), integrated with a novel algorithm for insulin bolus calculation. The aim of the ABC4D is to minimise high and low glucose excursions which are associated with the complications of diabetes including blindness, kidney failure, nerve damage and cardiovascular disease.

An interim analysis was conducted in Phase 4 after 25 participants completed the study (in line with the protocol) and it was agreed to stop the study at this stage. A further protocol amendment was approved by REC/MHRA to commence ABC4D phase 5 (different CT.gov number: NCT03963219).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Diagnosis of T1DM for > 1 year
* On MDI using a basal-bolus insulin regime
* Structured education in previous 3 years
* HbA1c ≤ 86mmol/mol
* No severe hypoglycaemia (defined as needing 3rd party assistance) in previous year

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Addison's Disease
* Gastroparesis
* Autonomic neuropathy
* Concomitant use of GLP-1 analogues and gliptins
* Visual impairment
* Reduced manual dexterity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Johnston, F.Med.Sci, Principal Investigator — Imperial College London; Nick Oliver, MRCP, Principal Investigator — Imperial College London; Monika Reddy, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This was not part of the approved protocol. Any peer-reviewed publications will be shared with the study participants and will be accessible to other researchers.

REFERENCES:
- [Derived] Reddy M, Pesl P, Xenou M, Toumazou C, Johnston D, Georgiou P, Herrero P, Oliver N. Clinical Safety and Feasibility of the Advanced Bolus Calculator for Type 1 Diabetes Based on Case-Based Reasoning: A 6-Week Nonrandomized Single-Arm Pilot Study. Diabetes Technol Ther. 2016 Aug;18(8):487-93. doi: 10.1089/dia.2015.0413. Epub 2016 May 19. PMID 27196358
- See also: Our research website — http://www3.imperial.ac.uk/bioinspiredtechnology/research/metabolic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From diabetes clinics
Groups:
- Phase 4 Intervention (ABC4D) & RT - CGM: Intervention (ABC4D) & Real-time continuous glucose monitoring over 6 months
- Phase 4 Control: Standard Bolus Calculator & RT-CGM: Control: standard bolus calculator & Real-time continuous glucose monitoring over 6 months
Period: Overall Study
Arm/Group | Phase 4 Intervention (ABC4D) & RT - CGM | Phase 4 Control: Standard Bolus Calculator & RT-CGM
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 4: Intervention (ABC4D) & RT - CGM: Intervention (ABC4D) & Real-time continuous glucose monitoring over 6 months
- Total: Total of all reporting groups
Arm/Group | Phase 4: Intervention (ABC4D) & RT - CGM | Phase 4 Control: Standard Bolus Calculator & RT-CGM | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (9.7) | 36.3 (14.1) | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Change in HbA1c
Time Frame: Baseline to 6 months
Measure: Median (Inter-Quartile Range); unit: mmol/mol
Groups:
- Intervention (ABC4D) & RT - CGM: Intervention (ABC4D) & Real-time continuous glucose monitoring
- Control: Standard Bolus Calculator & RT-CGM: Control: standard bolus calculator & Real-time continuous glucose monitoring
Arm/Group | Intervention (ABC4D) & RT - CGM | Control: Standard Bolus Calculator & RT-CGM
Number analyzed (Participants) | 13 | 12
mmol/mol | -5.0 [-11.5 to -4.0] | -3.0 [-10.3 to -0.8]
Statistical Analysis 1: Comparison: Intervention (ABC4D) & RT - CGM vs Control: Standard Bolus Calculator & RT-CGM; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage Time in Target Range
Description: Difference between baseline and 6-month endpoint.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Percentage
Groups:
- Phase 4 Intervention: ABC4D: ABC4D over 6 months in home setting
- Phase 4 Control: Standard Bolus Calculator: Standard bolus calculator for 6 months. real-time cGM in both groups.
Arm/Group | Phase 4 Intervention: ABC4D | Phase 4 Control: Standard Bolus Calculator
Number analyzed (Participants) | 13 | 12
Percentage | 0.9 [-1.4 to 3.6] | 0.0 [-3.6 to 3.8]

3. Secondary Outcome: Percentage Time in Hypoglycaemia
Description: Difference from baseline to 6-month endpoint.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Phase 4 Intervention: ABC4D | Phase 4 Control: Standard Bolus Calculator
Number analyzed (Participants) | 13 | 12
percentage | 0.5 [0.1 to 2.4] | -0.2 [-1.6 to 4.6]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Phase 4 Intervention & Control: Phase 4 Intervention (ABC4D)/Control group over 6 months
Arm/Group | Phase 4 Intervention & Control
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02053051/Prot_SAP_000.pdf